CLINICAL TRIAL: NCT02482350
Title: App-delivered Therapy for Arabic Readers With Hemianopic Alexia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University College London Hospitals (Other)
Responsible Party: Principal Investigator, Jenny Crinion, Dr, University College London Hospitals
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 150817
Record Dates: First submitted 2015-06-15; First posted 2015-06-26 (Estimated); Last update posted 2023-05-11 (Actual); Status verified 2023-05

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Reading Training (Experimental): A 3-months study design. There will be three distinct phases: base-line testing, reading training, and follow-up testing. T1-T7 indicate the 7 time-points at which we assess the following: reading speeds (word-per-minute), visual field test, visual search test, and Activities of Daily Living rating scale (T1: Day 1, Initial assessments; T2: Day 30, Pre-training assessments; T3: Day 60, During Reading Training (RT) after 5-hours; T4: During RT after 10-hours; T5: During RT after 15-hours; T6: During RT after 20-hour; T7: Day 90, Post-training assessments). Arabic reading patients with left-sided HA will receive app-delivered reading training in a single subject control based design for 1 month.
  Interventions: Behavioral: Reading Training

INTERVENTIONS:
Behavioral: Reading Training — Healthy subjects read moving (scrolling) text faster than static text. This type of text, also called "Times Square" presentation, induces a form of involuntary eye movement called optokinetic nystagmus (OKN) in the reader and, when used as part of a rehabilitation program, has been shown to improve subsequent reading performance of static text.

SUMMARY:
Hemianopia refers to compromised vision in one half of the visual field, in either one or both eyes. Hemianopic Alexia (HA) is a reading disorder related to such impairment, usually caused by stroke or head injury. In order to read, participants have to move their eyes along a line of text three to four times per second. Such eye movements are called saccades. One makes use of peripheral visual information to the right (if reading from left to right, e.g., in English) or to the left (if reading from right to left, e.g., in Arabic) of words. HA patients are deprived of much of this information. Patients with HA require far more saccades, which slows their reading significantly and often prevents them from reading efficiently for work or pleasure. It follows that the reading ability of those who read left-to-right would be compromised more by right-sided HA, and in those who read right-to-left by a left-sided HA. This study proposes to explore the rehabilitation of left-sided HA following stroke, in Arabic readers. An online treatment package has been developed in English (http://www.readright.ucl.ac.uk/). Currently, no assessment or treatment resources exist for the condition in right-to-left readers. The aim is to develop novel Arabic reading tests and rehabilitation material. The current project proposes to 1) translate this package into Arabic, 2) develop new Arabic reading test materials and 3) collect data from Arabic reading stroke patients in a Phase 2 clinical trial. The hope is to develop an effective, novel, and empirically supported reading treatment package for Arabic readers with HA.

DETAILED DESCRIPTION:
Background

Purpose and Experimental Design Reading a line of text is usually achieved by planning a series of saccades, which allow the eyes to jump from one word to another (reading scan-path). Arabic readers use peripheral visual information to the left of the word in order to plan their reading eye movements. Patients with HA are deprived of this information and compensate by creating inefficient reading scan-paths with many additional saccades, resulting in accurate but slow reading. Some patients abandon reading altogether, or lose their jobs because they cannot read fast enough.

Healthy subjects read moving (scrolling) text faster than static text. This type of text, also called "Times Square" presentation, induces a form of involuntary eye movement called optokinetic nystagmus (OKN) in the reader and, when used as part of a rehabilitation program, has been shown to improve subsequent reading performance of static text.

This study proposes to adapt these techniques for scrolling Arabic text, and to test them in Arabic-reading patients with left-sided HA. Rehabilitation material will be made available on the Internet (via an iPhone and/or iPad Application ('app')) for suitable subjects, in order to investigate whether patients benefit from using them outside of controlled trial conditions. During pre- and post-therapeutic intervention the investigators will record the following: reading speeds, visual field test scores, visual search test scores, eye-movements, and Activities of Daily Living scores. Length of time for which patients access rehabilitation material, will also be recorded.

This study will help determine the efficacy of Internet-based behavioural rehabilitation. It will also provide information as to: 1) how much improvement may be gained through this program, and 2) how much practice patients will likely require in order to improve their reading significantly.

Objectives

This study proposes:

1. Adapt and test reading rehabilitation techniques in patients with left-sided HA, using scrolling Arabic text;
2. Investigate whether patients benefit from using such material outside of controlled trial conditions.

Hypothesis

1. Patients will report a significant improvement in the speed at which they read static text (newspaper, books, letters, etc.) as a function of quality activity of daily living.
2. Patients will decrease the number of fixations (both progressive and regressive type saccades) when reading static text.

Methods Thirteen Arabic-reading patients with left-sided homonymous HA following stroke will be studied over a period of three months. A single-subject baseline control design will be employed. There will be a treatment-free interval before and after reading therapy. Baseline assessments of visual fields, eye movement performance during text reading, text reading speed, and visual search performance will be carried out pre-intervention. Behavioural assessments will be repeated immediately following every five hours of therapy, and during follow-up. Patients will determine how long to wait between testing points, as they will differ in reading speeds.

Patients meeting the study criteria will be identified through Dr. Alex Leff's Alexia clinic at the National Hospital for Neurology and Neurosurgery, University College London Hospital (UCLH), as well as through formal collaboration with the neuropsychology department at Wellington Hospital. In addition, patients will be given the option to join the study when downloading the reading therapy app from the Apple iTunes store. An online consent form will be included in the registration. The aim is to recruit at least thirteen patients to this study over the following three years.

Thirteen healthy age-matched Arabic reading controls will be recruited from a variety of sources, including relatives and friends of patients. Controls will undergo the same assessment as patients, but will be assessed only once. They will not undergo the reading therapy.

Consent Initially, both the information sheet and consent forms will be delivered in hard copy (written in both Arabic and English). When the application has been developed, pilot study will be conducted. Participants will complete online consent forms, and will be required to click certain key boxes to confirm that they have read or listened to, and understood, the information.

Risks, Burdens, and Benefits:

Benefits. App-delivered reading therapy has never before been available as a rehabilitation package for Arabic reading patients with HA. The app may be used as stand-alone self-help reading therapy, or as part of formal speech-language therapy. Additional benefits include real-time activity monitoring, tracking of treatment progress, personalised feedback and motivation support, portability and flexibility of use, and the potential to improve with practice.

Risks/Burdens. This will be the first study in patients with left-sided HA using scrolling Arabic text. Thus there is little literature to guide the study. In order to maximize its potential, the investigators will adapt the established English-reading treatment approach used for patients with right-sided HA. There is no way of predicting how many patients will use the application. Some participants may not meet the study criteria. In addition, the patients themselves will manage their use of the application. There is therefore an inherent risk of their not accessing the rehabilitation materials for the required period of time, and not entering the data correctly.

Data Collection

Participants will be required to enter the following data in order to gain full access to the rehabilitation material:

Data to be collected on App-based patients

1. A unique login, created by themselves. (This does not have to be their real name.) This will ensure that each time they access the application; their data is collected under their name.
2. Their email address (optional), for use only if they forget their login details.
3. The extent and side of their hemianopia. If they have not had this test performed by their own doctor or optometrist, a section of this application provides self-testing.
4. A test of their reading speed. This will be self-administered. Participants will time themselves (a timer on the application will be activated by the touch screen) reading a standard text aloud. Their text reading speed will be calculated and feedback to them. Participants may check or recheck this at various times during the study.
5. A test of their performance on a visual search test. This will be self-administered. Participants will be tested on their accuracy and speed when finding objects on a section of the application. Their performance scores will be calculated and feedback to them. Participants may check or recheck this at various times during the study.
6. Participants will rate themselves on their ability to perform activities of daily living (ADLs) as a measure of their functional status in regards to their reading impairment. Their scores will be calculated but not feedback to them.

Other optional fields, which may prove useful in data analysis if enough subjects complete them will include:

1. The cause of their hemianopia. (This is usually stroke or head injury, but a free text option will be provided.)
2. How much reading they can manage with their hemianopia
3. Whether their hemianopia has caused them to change or loose their employment

Participants will access the app and enter all personal data themselves. The only data we will collect that is not directly controlled by the participants is the amount of time they access the rehabilitation materials and their logon identification. The latter will ensure that the same participant is not logging on to the application under multiple names.

Rehabilitation materials used in the app-based reading training The rehabilitation materials will consist simply of chapters of text, which scroll from left-to-right: that is, from the blind visual field of the participants to their normal visual field. The texts will be sourced from books out of copyright, freely available on the Internet. The aim is to provide streaming text from other websites, such as news, current affairs etc. The participant may control the speed at which the text scrolls. Participants will be advised to practice the reading therapy on most days and to aim for 20 to 40 minutes per day. They will also be asked to test their reading speeds every time they complete five hours of rehabilitation. Subjects will be prompted to check their reading speeds after every five hours of exposure to therapy. If they choose not to record any of this data, their access to the rehabilitation materials will not be affected.

Data to be collected on Face-to-Face patients Patients with HA adopt an inefficient reading strategy to compensate for their visual impairment on the hemianopic side. Therefore, we want to compare the patients' reading scan-paths to those generated by healthy controls reading the same static passages. We will be recording eye movements of participants as they read 10 passages using an eye-tracking device. A between groups statistical analysis will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Participants must:

  1. Have a right-sided hemispheric stroke, tumor or head injury
  2. Demonstrate a fixed left visual field homonymous deficit as defined by missing one or more stimuli on the automated visual field test developed for the application
  3. Have a baseline text reading speed of more than 40 words per minute
  4. Have been Arabic readers premorbidly

Exclusion Criteria:

* Patients presenting:

  1. impaired speech production, speech comprehension or writing (to rule out those with central alexia)
  2. a premorbid history of neurological or psychiatric illness
  3. a baseline text reading speed of less than 40 words per minute (to exclude patients with pure alexia) will be excluded from the study

Ages: 26 Years to 81 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2015-07; Primary Completion 2018-09 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
Improvement of reading speed | 1 month
  Average total reading time will be calculated in words per minute (wpm) using descriptive statistics in IBM SPSS.

SECONDARY OUTCOMES:
Patients will report improvement in static text reading (newspapers, books, letters, etc.) as a function of quality activity of daily living. | 2 months
  Participants will rate themselves on their ability to perform activities of daily living (ADLs) as a measure of their functional status in regards to their reading impairment.
Decrease in the number of fixations | 1 month
  Fixation: maintaining visual gaze on a single location
Decrease in average fixation durations | 1 month
  Fixation duration: length of fixational pauses during reading

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer T Crinion, PhD, Principal Investigator — Institute of Cognitive Neuroscience
Locations (1):
- The Wellington Hospital, London, United Kingdom